CLINICAL TRIAL: NCT05370131
Title: The Effect of An Avatar-Based Education Program Developed For The Care Of Children With Ventriculoperitoneal Shunts On Shunt Complications And Parents' Knowledge And Care Skills: A Multicenter Randomized Controlled Trial
Brief Title: The Effect of an Avatar-Based Education Program on Shunt Complications and Parents' Knowledge and Care Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Mustafa Volkan DÜZGÜN, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KAEK-98; 221S685 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2022-04-03; First posted 2022-05-11 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Developing the ABEP-H; Determining the Effect of ABEP-H
Keywords: hydrocephalus; avatar-based education program; pediatric nursing; shunt complication; parents' knowledge and care skill
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatar-Based Education Program in Hydrocephalus (ABEP-H) (Experimental): The avatar-based education program in hydrocephalus (ABEP-H) aimed to help parents acquire the knowledge and develop the skills necessary for the care of hydrocephalus children with VP shunts and prevent shunt infection and dysfunction. The intervention group participants will be sent usernames and passwords they can change by accessing their profiles. The main researcher will show them how to log into the program and use it on their phones and computers. This interview will take about 40 minutes. Afterward, they are expected to use the program for six months on a regular basis. Their login frequency and duration will be monitored. After six months, they will be asked to fill out the System Usability Scale (SUS). Moreover, each participant will be phoned once every two weeks as a reminder.
  Interventions: Other: Avatar-Based Education Program in Hydrocephalus (ABEP-H)
- Control Group (No Intervention): The control group will receive the standard care procedures of the hospital.

INTERVENTIONS:
Other: Avatar-Based Education Program in Hydrocephalus (ABEP-H) — The avatar-based education program in hydrocephalus (ABEP-H) aimed to help parents acquire the knowledge and develop the skills necessary for the care of hydrocephalus children with VP shunts and prevent shunt infection and dysfunction.
  Arms: Avatar-Based Education Program in Hydrocephalus (ABEP-H)

SUMMARY:
Hydrocephalus is a common childhood neurosurgical disease. Ventriculoperitoneal (VP) shunt is usually used in the treatment of hydrocephalus. However, VP shunt may have some complications. In developed countries, the incidence of hydrocephalus is 1 per 1000 live births. In developing countries, it is 3-4 per 1000 live births. A multidisciplinary approach is important in the treatment and care of hydrocephalus. Parents need guidance and training for hydrocephalus treatment and care. Nurses should help parents solve all care-related problems. Technology-based nursing interventions have become popular in recent years because they make life easier for children with chronic diseases and their parents who should avoid non-emergency hospital visits during the COVID-19 pandemic. Investigators need innovative and interactive technology-based interventions to provide patients and their parents with the knowledge and skills necessary to manage chronic diseases. This study also focused on an avatar-based education program because avatars are interactive icons that provide intrinsic and extrinsic motivation for parents. Therefore Investigators develop an Avatar-based education program in Hydrocephalus (ABEP-H) and prove its effectiveness in reducing shunt complications and helping parents acquire the knowledge and develop the skills necessary for the care of their children with hydrocephalus.

DETAILED DESCRIPTION:
Ventriculoperitoneal (VP) shunt is usually used in the treatment of hydrocephalus. However, VP shunt may have some complications. Children with shunts need good primary care.

There have been significant advances in science and technology in recent years. Therefore, education programs for patients and their parents also involve technology. The new face of technology in patient education is avatar-based education programs used to manage chronic diseases (cancer, diabetes, depression, etc.). However, this technology is underutilized in the training of pediatric patients. Therefore, this study will present a randomized controlled trial protocol to develop an avatar-based education program and determine its effect on shunt complications and parents' knowledge and care skills (ABEP-H).

The ABEP-H protocol adopted a single-blind, pretest-posttest, parallel-group (1:1 ratio), follow-up, multicenter randomized controlled experimental design. The intervention group will attend the ABEP-H for six months. Each intervention group participant will be phoned once every two weeks as a reminder. Data will be collected in the first, third, and sixth months.

The ABEP-H protocol will be based on the template for intervention description and replication (TIDieR) guideline and checklist. The protocol is designed according to the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT). Randomized controlled trials (RCTs) are reported based on the Consolidated Standards of Reporting Trials (CONSORT).

ELIGIBILITY:
Inclusion Criteria:

* Having a child with a VP shunt in the past six months
* No shunt infection
* Having a smartphone and mobile Internet access
* Speaking Turkish
* Understanding what is read and said
* Executing commands

Exclusion Criteria:

* Not using the ABEP-H actively

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
VP Shunt Complication Follow-up List (VP-CFL) | 1. month
  The VP Shunt Complication Follow-up List (VP-CFL) was based on a literature review conducted by the researchers. It consists of 24 parameters about shunt infection and dysfunction. These data will be provided from the patient file. The researcher will collect data on the other parameters during routine consultations and physical examinations. The follow-up of shunt complications in children will be done through this list.
VP Shunt Complication Follow-up List (VP-CFL) | 3. months
  The VP Shunt Complication Follow-up List (VP-CFL) was based on a literature review conducted by the researchers. It consists of 24 parameters about shunt infection and dysfunction. These data will be provided from the patient file. The researcher will collect data on the other parameters during routine consultations and physical examinations. The follow-up of shunt complications in children will be done through this list.
VP Shunt Complication Follow-up List (VP-CFL) | 6. months
  The VP Shunt Complication Follow-up List (VP-CFL) was based on a literature review conducted by the researchers. It consists of 24 parameters about shunt infection and dysfunction. These data will be provided from the patient file. The researcher will collect data on the other parameters during routine consultations and physical examinations. The follow-up of shunt complications in children will be done through this list.
Hydrocephalus Knowledge and Care Skills Self-Assessment Scale | At the beginning of the research
  The researchers are developing the Hydrocephalus Knowledge and Care Skills Self-Assessment Scale (HKCSSAS). It is aimed to measure the knowledge and care skills of parents.The results of the pilot study showed that the scale was valid and reliable.
Hydrocephalus Knowledge and Care Skills Self-Assessment Scale | 6. months
  The researchers are developing the Hydrocephalus Knowledge and Care Skills Self-Assessment Scale (HKCSSAS). It is aimed to measure the knowledge and care skills of parents.The results of the pilot study showed that the scale was valid and reliable.

SECONDARY OUTCOMES:
Child and Parent Descriptive Questionnaire | At the beginning of the research
  The Child and Parent Descriptive Questionnaire (CPDQ) was based on a literature review conducted by the researchers. It consists of two parts. The first part consists of 10 items on children's sociodemographic characteristics and hydrocephalus. The second part consists of 13 items on parents' sociodemographic characteristics.
System Usability Scale (SUS) | 6. Months
  The System Usability Scale (SUS) was developed by John Brooke and adapted to Turkish by Demirkol and Şeneler to measure the usability of products and services (hardware, software, mobile devices, websites, apps, etc.). The instrument consists of ten items rated on a five-point Likert-type scale (0: strongly disagree, 1: disagree, 2: undecided, 3: agree, 4: strongly agree). Five items (2, 4, 6, 8, and 10) are reverse scored. Each score is multiplied by 2.5 to convert to a scale of 0 to 100, where 100 represents the best possible usability.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül ISLER DALGIC, Prof, Study Director — Akdeniz University; Mehmet Saim KAZAN, Prof, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will not be shared for the purpose of confidentiality and protection of personal data.